CLINICAL TRIAL: NCT05112731
Title: Action of Glycation and Inflammation in Operative Ischemic Heart Disease
Brief Title: Role of Glycation and Inflammation in Acute Ischemic Heart Disease
Acronym: AGLIANICO
Status: Terminated | Type: Observational
Why Stopped: Missing enrollment at study centre
Sponsor: GEK Srl (Industry)
Collaborators: Istituto Clinico Città Studi (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021AGLIANICO
Record Dates: First submitted 2021-10-20; First posted 2021-11-09 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction; Glycation End Products, Advanced; Inflammation; Heart Injuries; Heart Inflammation
Keywords: AGEs; BAFF; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Heart Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- First Ischemic Cardiac Event: Measurement of BAFF and MGO at hospitalization (before reperfusion) and after 3 months during follow-up
  Interventions: Diagnostic Test: BAFF and MGO

INTERVENTIONS:
Diagnostic Test: BAFF and MGO — measurement of BAFF and MGO levels before reperfusion and after 3 months

SUMMARY:
This study requires the consecutive enrollment of 60 patients following the first event of acute myocardial infarction, evaluating B-Cell Activating Factor (BAFF) and methylglyoxal (MGO) levels in the acute setting (pre-reperfusion) and 3 months after reperfusion.

DETAILED DESCRIPTION:
This study requires the consecutive enrollment of 60 patients at admission for first acute myocardial infarction. At enrollment, before reperfusion, a blood sample is obtained to measure B-Cell Activating Factor (BAFF) and methylglyoxal (MGO) levels in the acute setting. This measure is then repeated at follow-up visit 3 months after reperfusion. The aim of the study is to identify specific subsets of patients and evaluate biomarkers variations.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization for first myocardial infarction (STEMI or NSTEMI)
* age between 18 and 80

Exclusion Criteria:

* uncompensated T2DM (HbA1c >53mmol/mol)
* use of anti-CD20 treatment
* chronic anti-inflammatory treatment for autoimmune disease (i.e. DMARDs, high dose FANS, cortisonic drugs)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 consecutive patients admitted in the ED for first myocardial infarction who meet eligibility criteria
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Identification of Inflammatory Biomarkers (BAFF) linked to ischemic event and outcome | Day 0
  elevation of BAFF levels
Identification of Glycation Biomarkers (MGO) linked to ischemic event and outcome | Day 0
  elevation of MGO levels

SECONDARY OUTCOMES:
Identification of biomarkers variations (BAFF) complications and outcome | After 3 months
  variation of BAFF from baseline
Identification of biomarkers variations (MGO) complications and outcome | After 3 months
  variation of MGO from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bianchi, MD, Principal Investigator — Istituto Clinico Città Studi; Altin Palloshi, MD, Principal Investigator — Istituto Clinico Città Studi
Locations (1):
- Istituto Clinico Città Studi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evans JDW, Dobbin SJH, Pettit SJ, Di Angelantonio E, Willeit P. High-Sensitivity Cardiac Troponin and New-Onset Heart Failure: A Systematic Review and Meta-Analysis of 67,063 Patients With 4,165 Incident Heart Failure Events. JACC Heart Fail. 2018 Mar;6(3):187-197. doi: 10.1016/j.jchf.2017.11.003. Epub 2018 Jan 10. PMID 29331272
- [Background] Mariathas M, Allan R, Ramamoorthy S, Olechowski B, Hinton J, Azor M, Nicholas Z, Calver A, Corbett S, Mahmoudi M, Rawlins J, Simpson I, Wilkinson J, Kwok CS, Cook P, Mamas MA, Curzen N. True 99th centile of high sensitivity cardiac troponin for hospital patients: prospective, observational cohort study. BMJ. 2019 Mar 13;364:l729. doi: 10.1136/bmj.l729. PMID 30867154
- [Background] Francis Stuart SD, De Jesus NM, Lindsey ML, Ripplinger CM. The crossroads of inflammation, fibrosis, and arrhythmia following myocardial infarction. J Mol Cell Cardiol. 2016 Feb;91:114-22. doi: 10.1016/j.yjmcc.2015.12.024. Epub 2015 Dec 29. PMID 26739214
- [Background] Zouggari Y, Ait-Oufella H, Bonnin P, Simon T, Sage AP, Guerin C, Vilar J, Caligiuri G, Tsiantoulas D, Laurans L, Dumeau E, Kotti S, Bruneval P, Charo IF, Binder CJ, Danchin N, Tedgui A, Tedder TF, Silvestre JS, Mallat Z. B lymphocytes trigger monocyte mobilization and impair heart function after acute myocardial infarction. Nat Med. 2013 Oct;19(10):1273-80. doi: 10.1038/nm.3284. Epub 2013 Sep 15. PMID 24037091
- [Background] Akhand AA, Hossain K, Mitsui H, Kato M, Miyata T, Inagi R, Du J, Takeda K, Kawamoto Y, Suzuki H, Kurokawa K, Nakashima I. Glyoxal and methylglyoxal trigger distinct signals for map family kinases and caspase activation in human endothelial cells. Free Radic Biol Med. 2001 Jul 1;31(1):20-30. doi: 10.1016/s0891-5849(01)00550-0. PMID 11425486
- [Background] Khan MA, Schultz S, Othman A, Fleming T, Lebron-Galan R, Rades D, Clemente D, Nawroth PP, Schwaninger M. Hyperglycemia in Stroke Impairs Polarization of Monocytes/Macrophages to a Protective Noninflammatory Cell Type. J Neurosci. 2016 Sep 7;36(36):9313-25. doi: 10.1523/JNEUROSCI.0473-16.2016. PMID 27605608
- [Background] Blackburn NJR, Vulesevic B, McNeill B, Cimenci CE, Ahmadi A, Gonzalez-Gomez M, Ostojic A, Zhong Z, Brownlee M, Beisswenger PJ, Milne RW, Suuronen EJ. Methylglyoxal-derived advanced glycation end products contribute to negative cardiac remodeling and dysfunction post-myocardial infarction. Basic Res Cardiol. 2017 Sep 1;112(5):57. doi: 10.1007/s00395-017-0646-x. PMID 28864889